CLINICAL TRIAL: NCT03837964
Title: Relative Bioavailability of BI 1291583 Following Oral Administration Under Fed and Fasted Conditions in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Study)
Brief Title: A Study to Test How Food Influences the Amount of BI 1291583 in the Blood of Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1397-0008; 2018-001274-14 (EudraCT Number)
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment T (Experimental): Fed
  Interventions: Drug: BI 1291583
- Treatment R (Experimental): Fasted
  Interventions: Drug: BI 1291583

INTERVENTIONS:
Drug: BI 1291583 — Tablet
  Other Names: Verducatib

SUMMARY:
To assess the effect of food on the pharmacokinetics of an oral tablet formulation of BI 1291583, by investigating the relative bioavailability following single dose administration under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good clinical practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR), or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are greater than 450 ms, if confirmed by a second Electrocardiogram (ECG) recording) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 1291583 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Within 3 hours (h) before and 0.5, 1, 2, 4, 5, 6, 7, 8, 10, 12, 14, 24, 34, 48, 72, 96, 120, 168, 216, 264 hours after drug administration
  Area under the concentration-time curve of BI 1291583 in plasma over the time interval from 0 to the last quantifiable data point.
Maximum measured concentration of BI 1291583 in plasma (Cmax) | Within 3 hours (h) before and 0.5, 1, 2, 4, 5, 6, 7, 8, 10, 12, 14, 24, 34, 48, 72, 96, 120, 168, 216, 264 hours after drug administration
  Maximum measured concentration of BI 1291583 in plasma

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 1291583 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) | Within 3 hours (h) before and 0.5, 1, 2, 4, 5, 6, 7, 8, 10, 12, 14, 24, 34, 48, 72, 96, 120, 168, 216, 264 hours after drug administration
  AUC0-inf represents the area under the concentration-time curve of BI 1291583 in plasma over the time interval from 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/